CLINICAL TRIAL: NCT07371130
Title: Evaluation of Low-Intensity Therapeutic Wavelength Nanotechnology Devices in Alveolar Preservation: A Clinical Trial
Brief Title: Therapeutic Wavelength Nanotechnology Devices in Alveolar Preservation
Acronym: APnanotecnolog
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Dr, University of Bari Aldo Moro
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AlveolarPreservation
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Tooth Avulsion; Tooth Crown Fracture
Keywords: alveolar ridge preservation; alveolar preservation; bone loss; bone preservation
MeSH Terms: conditions — Tooth Avulsion; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Alveolar Preservation (Active Comparator): The socket is filled with a xenogeneic bone graft enriched with hyaluronic acid and dermal membrane
  Interventions: Procedure: Socket Preservation
- therapeutic wavelengths Alveolar Preservation (Experimental): Therapeutic wavelengths are applied as part of the alveolar preservation protocol. The extraction socket is filled with a xenogeneic bone graft enriched with hyaluronic acid and subsequently covered with a dermal membrane to support healing and tissue regeneration.
  Interventions: Procedure: Socket Preservation

INTERVENTIONS:
Procedure: Socket Preservation — After atraumatic tooth extraction, the socket is filled with a xenogeneic bone graft enriched with hyaluronic acid, which enhances biological activity by promoting angiogenesis, cell migration, and early wound healing. The grafted site is then covered with a dermal matrix membrane, providing mechanical protection, stabilization of the biomaterial, and guided tissue regeneration.

SUMMARY:
After tooth extraction, a progressive alveolar bone resorption is observed. Alveolar ridge preservation consists of placing a biomaterial within the extraction socket and covering it with a membrane.

This procedure helps limit physiological bone resorption, making the soft and hard tissue profile of the edentulous site more prosthetically favorable.

DETAILED DESCRIPTION:
After tooth extraction, a progressive remodeling process occurs that is often associated with significant alveolar bone resorption, particularly in sites with compromised bony walls. Alveolar ridge preservation is a surgical procedure aimed at minimizing this physiological resorption by placing grafting materials within the extraction socket and protecting them with a barrier membrane.

In the present protocol, the socket is filled with a xenogeneic bone graft enriched with hyaluronic acid, which enhances biological activity by promoting angiogenesis, cell migration, and early wound healing. The grafted site is then covered with a dermal matrix membrane, providing mechanical protection, stabilization of the biomaterial, and guided tissue regeneration.

In one study group, in addition to the surgical procedure, postoperative biostimulation using low-intensity photonic nanotechnology is applied. This adjunctive therapy is intended to enhance cellular metabolism, modulate inflammation, and accelerate both soft and hard tissue healing. The combined approach aims to preserve alveolar volume more effectively, improve the quality of regenerated tissues, and create a more favorable prosthetic environment for subsequent implant rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults in good general health
* Indication for tooth extraction in sites planned for delayed implant placement
* Inability to place immediate post-extraction implants due to insufficient residual bone to ensure primary stability
* Extraction sockets presenting absence of the buccal (vestibular) bone wall
* Signed informed consent

Exclusion Criteria:

* Systemic conditions affecting bone healing
* Uncontrolled periodontal disease
* Smoking >10 cigarettes/day
* Pregnancy or lactation
* Use of medications interfering with bone metabolism

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
VAS | 1 day , 3 days , 7 days ,14 days
  Postoperative pain assessment using the Visual Analog Scale (VAS) (1-10)
Analgesic consumption | 7 days
  recorded as the number of ibuprofen 400 mg tablets taken

SECONDARY OUTCOMES:
Histological Evaluation | 4- 6 month
  * Prior to implant placement, a CBCT scan will be performed to assess alveolar bone volume and morphology.
  * During implant site preparation, a bone core biopsy will be harvested using a trephine bur.
  * The bone sample will undergo histological and histomorphometric analysis to evaluate:
    * New bone formation
    * Residual graft material
    * Connective tissue percentage

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe D'Albis, Dr., Principal Investigator — University of Bari Aldo Moro; Domenico Patarino, Dr., Principal Investigator — Private Practice; Saverio Capodiferro, Prof. Dr., Study Director — University of Bari Aldo Moro